## Official Title: IVY: Intervention for Victimized Youth

NCT Number: NCT06631274

**Document Date: October 18, 2024** 

**Analytic Plan** 

## **Analytic Plan**

Statistical analyses included three steps. First, missing data occurred only on items measuring social support. Little's test was used to examine the tenability of the assumption of missing completely at random. Second, the mean scores across items in each scale/subscale were computed to represent each intermediate and distal outcome. Third, a series of one-way repeated measures ANOVAs was conducted to examine the impact of intervention, in which participation in the intervention (treatment vs. control) was used as the between-subject factor and time points (time 1 and time 2) was used as the within-subject factor. In addition to significance test for main effect of group, main effect of time, and the interaction effect between time and group, Hedges' g was computed to indicate effect size, where values of 0.2, 0.5, and 0.8 indicate a small, medium, and large effect respectively.